CLINICAL TRIAL: NCT04682509
Title: A Single-center Pilot Study Evaluating a Preemptive Short Course of Glecaprevir/Pibrentasvir in Hepatitis C Positive to Negative Kidney Transplantation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-01386
Record Dates: First submitted 2020-12-22; First posted 2020-12-23 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: ESRD
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): All study subjects will receive glecaprevir/pibrentasvir (Mavyret®) 300/120 mg orally x 14 days, starting on POD 0 prior to transplantation of the HCV positive kidney. If HCV RNA is detectable after 2 weeks of therapy, Mavyret® will be continued to complete a full course of 8 weeks per standard of care. Safety monitoring and frequent surveillance for HCV viremia will occur for all subjects throughout the duration of the study. The kidney transplantation procedure and routine post-transplant management will be performed per standard of care.
  Interventions: Drug: Glecaprevir/pibrentasvir

INTERVENTIONS:
Drug: Glecaprevir/pibrentasvir — Manufacturer is AbbVie, Inc., North Chicago, IL Mavyret® is commercially available and FDA approved for the treatment of HCV genotype 1, 2, 3, 4, 5, or 6 infection in patients without cirrhosis or with compensated cirrhosis and also for the treatment of adult patients with HCV genotype 1 infection who previously have been treated with a regimen containing an HCV NS5A inhibitor or an NS3/4A protease inhibitor. An immediate release bilayer oral tablet containing a fixed-dose combination of 100 mg of glecaprevir and 40 mg of pibrentasvir. The daily dose of glecaprevir/pibrentasvir used will be the standard FDA approved dose: 3 tablets taken once daily (total daily dose: glecaprevir 300 mg and pibrentasvir 120 mg).
  Other Names: Mavyret

SUMMARY:
The purpose of this research study is to evaluate the feasibility of a 2 week course of glecaprevir/pibrentasvir (Mavyret) starting immediately prior to transplantation to treat hepatitis C virus (HCV) in kidney transplant recipients who receive a kidney from a donor with HCV.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-center, pilot study. The patient population will include 20 patients who are on the kidney transplant waitlist at NYU Langone Health, are hepatitis C virus (HCV) negative, are willing to accept an organ from an HCV positive donor, and consent to participate in this trial. Study subjects will receive a kidney transplant from a deceased donor who tested positive for HCV as confirmed by nucleic acid amplification testing (NAT) per standard of care. All study subjects will receive a two week course of preemptive therapy with glecaprevir/pibrentasvir (Mavyret®), starting on postoperative day (POD) 0 prior to the transplant. If HCV RNA is undetectable after 2 weeks of therapy, Mavyret will be discontinued and study subjects will be followed with an intensive HCV monitoring protocol. If HCV RNA is detectable after 2 weeks of therapy, Mavyret will be continued to complete a full course of 8 weeks per standard of care. All patients will undergo close monitoring and surveillance for HCV viremia post-transplant to ensure that sustained virologic response (SVR) is achieved.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Listed for kidney transplantation at NYU Langone Health and willing to accept HCV positive donor organs
* Able to complete routine post-transplant visits and study visits for a minimum of 1 year after transplantation
* Women of childbearing potential must agree to use birth control in accordance with Mycophenolate Risk Evaluation and Mitigation Stategy (REMS) after transplant due to increased risk of birth defects and/or miscarriage
* Both men and women must agree to use at least one barrier method of contraception after transplant to prevent any secretion exchange
* Able and willing to provide informed consent
* Receive an organ offer for a kidney from a deceased donor that:
* Is HCV NAT positive
* Meets all standard criteria for organ acceptability at NYU Langone Transplant Institute

Exclusion Criteria:

* HCV RNA positive or history of previously treated HCV
* Evidence of active hepatitis B infection or on active antiviral treatment of HBV
* HIV positivity
* Pregnant or nursing (lactacting) women
* Current use of atazanavir or rifampin
* Known hypersensitivity to glecaprevir and/or pibrentasvir
* Current or history of decompensated liver disease
* Recipients of dual organs (i.e. simultaneous liver and kidney transplant, simultaneous kidney and pancreas transplant, or simultaneous heart and kidney transplant)
* Receive an organ offer for a kidney from a deceased donor that is:
* Confirmed HIV positive
* Confirmed HBV positive (positive hepatitis B surface antigen, and/or detectable hepatitis B virus DNA)
* Known to have previously failed DAA therapy for treatment for HCV
* HCV antibody positive, but NAT negative

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Change in the Percentage of Incidence of sustained clearance of HCV (cure) 12 weeks after treatment of viremia | Visit 2 (Day 1) , Visit 3 (Day 3) , Visit 4 (Day 7), Visit 5 (Day 13), Visit 16 (Day 365)
  Measured in percentage of patients with SVR after treatment for HCV after kidney transplant. SVR will be defined as the absence of detectable HCV RNA Quantitative (PCR) testing 12 weeks after the completion of the treatment course.

SECONDARY OUTCOMES:
Percentage of Overall patient and graft survival at 1 year post-transplant | Visit 1 (Day 0), Visit 16 (Day 365)
  Patients will have regular follow-up as standard-of-care for all kidney transplant recipients. Patients' survival will be readily apparent. Furthermore, all deaths of transplant recipients and allograft losses within the first year of transplant are required to be reported to UNOS. Survival rates will be reported as a percentage.
Change in the Allograft function | Visit 1 (Day 0), Visit 16 (Day 365)
  This parameter is being used to measure overall graft function and will be described using the median value at 1 year post transplant for the cohort. All transplant recipients will have regular follow-up as standard-of-care and eGFR will be calculated using the MDRD equation.
Percentage of Incidence and grade of biopsy-proven rejection | Visit 1 (Day 0), Visit 16 (Day 365)
  All transplant recipients will have regular follow-up as routine clinical care and as such, will receive for cause biopsies per standard of care if there is a clinical suspicion of rejection. Biopsies will be read by a renal pathologist per standard of care and reported in the EPIC system. The incidence of rejection will be calculated as a percentage of the patients with diagnosed rejection on biopsy within 1 year of transplant.
Time course to transplantation (median) | Screening vist, Visit 1 (Day 0)
  Time to transplantation will be measured from the time of listing (recorded in EPIC) to time of transplant and also time from written acknowledgment of willingness to participate in the trial to time of transplant.
Percentage of Incidence HCV viremia post-transplant and after 2 weeks of treatment | Visit 1 (Day 0), Visit 5 (Day 13), Visit 16 (Day 365)
  Measuring serial HCV RNA Quantitative (PCR) starting immediately after transplant and continued throughout the duration of the study. A patient will be considered to be viremic when a post-transplant HCV RNA Quantitative (PCR) test is positive. The incidence of viremia after transplant will be calculated as the percent of the patients transplanted with an HCV-positive donor who subsequently developed HCV viremia (detected by RNA Quantitative (PCR) testing). The incidence of viremia after two weeks of treatment will be calculated as the percentage of the patients with detectable HCV viremia (detected by RNA Quantitative (PCR) testing) after completing 2 weeks of treatment with glecaprevir/pibrentasvir and therefore require continuation of therapy to complete an 8 week course
Time course of exposure to development of clinically detectable viremia in those who develop viremia | Visit 1 (Day 0) to Visit 16 (Days 364)
  Measuring serial HCV RNA Quantitative (PCR) starting immediately after transplant and continued throughout the duration of the study to find the median time to viremia with standard deviations. If the HCV RNA Quantitative (PCR) test is positive at any time point, we will calculate the time from transplant to detectable HCV RNA Quantitative (PCR).
Time course of clearance of viremia after treatment initiation | Visit 1 (Day 0) to Visit 16 (Days 364)
  Measuring serial HCV RNA Quantitative (PCR) starting immediately after transplant and continued throughout the duration of the study to find the median time to clearance with standard deviations. If the HCV RNA Quantitative (PCR) test is positive at any time point, we will calculate the time to documented clearance as indicated by an undetectable HCV RNA Quantitative (PCR),
Percentage of Incidence of treatment failure/treatment resistant strains of HCV | Visit 1 (Day 0), Visit 5 (Day 13), Visit 9 (Day 56)
  If SVR12 is not achieved with either a 2 week or 8 week course of glecaprevir/pibrentasvir, it will be considered a treatment failure and resistance testing will be performed. The incidence will be reported as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Lonze, MD, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This is a single center pilot study. Data will be available once published.